CLINICAL TRIAL: NCT04630262
Title: Multi-Center Clinical Investigation of the ATTUNE® Cementless Fixed Bearing Tibial Base and Cementless Patella Implants in Total Knee Arthroplasty
Brief Title: ATTUNE Cementless FB Tibial Base Clinical Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was unfunded.
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSJ_2019_05
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Post-traumatic arthritis; Failed total knee; Knee; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: ATTUNE Cementless Fixed Bearing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ATTUNE Cementless CR Fixed Bearing (Active Comparator): Subjects enrolled who undergo TKA with the ATTUNE Cementless Fixed Bearing Cruciate Retaining Configuration.
  Interventions: Device: ATTUNE Cementless CR Fixed Bearing
- ATTUNE Cementless PS Fixed Bearing (Active Comparator): Subjects enrolled who undergo TKA with the ATTUNE Cementless Fixed Bearing Posterior Stabilizing Configuration.
  Interventions: Device: ATTUNE Cementless PS Fixed Bearing

INTERVENTIONS:
Device: ATTUNE Cementless CR Fixed Bearing — Subjects Implanted with the ATTUNE Cementless Femoral, Cementless Tibia, and CR or (Medial Stabilized) MS Tibial Insert.
  Arms: ATTUNE Cementless CR Fixed Bearing
Device: ATTUNE Cementless PS Fixed Bearing — Subjects Implanted with the ATTUNE Cementless Femoral, Cementless Tibia, and PS Tibial Insert.
  Arms: ATTUNE Cementless PS Fixed Bearing

SUMMARY:
This is a prospective, multi-center, non-randomized, single arm observational study. The primary objective of this clinical investigation is to evaluate functional responder rates with an objective performance criteria (OPC) of 85% as measured by the KOOS questionnaire for the first 225 tibia (CR FB and PS FB combined) implanted with the ATTUNE Cementless FB tray (primary and revision procedures) and will be analyzed when these patients have passed the 1 year preferred post-op window.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to evaluate functional responder rates with an objective performance criteria (OPC) of 85% as measured by the KOOS questionnaire for the first 225 tibia (CR FB and PS FB combined) implanted with the ATTUNE Cementless FB tray (primary and revision procedures) and will be analyzed when these patients have passed the 1 year preferred post-op window. Study success will be determined using the primary TKA (CR FB and PS FB combined) analysis group.

The secondary objectives of this study are to establish the surgical effectiveness of the ATTUNE Cementless Tibial Base by evaluating type and frequency of Adverse Events and Device Deficiencies, functional responder rates with an objective performance criteria (OPC) of 85% as measured by the KOOS questionnaire for all subjects (CR FB and PS FB combined) at the 1-year timepoint, the change from preoperative baseline to the 6-week, 6-month, 1-year, 2-year and 5-year timepoints in functional outcomes and quality of life assessments, as measured using additional patient reported outcomes measures (PROMS), implant survivorship of the ATTUNE Cementless FB Tibial base using Kaplan-Meier survival analysis at 1, 2 and 5-year timepoints, and investigator-conducted radiographic analysis of the tibial and patellar components at 6 weeks/6 months 1, 2 and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and between the ages of 22 and 80 years at the time of consent, inclusive.
2. Subject has a severely painful knee and/or impaired knee function resulting from osteoarthritis, post-traumatic arthritis, or a failed previous implant provided that adequate bone is present.
3. Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor.
4. Subject is currently not bedridden.
5. Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.
6. Subject is able to read and comprehend the Informed Consent Document as well as complete the required PROMs in either English or one of the available translations.

Exclusion Criteria:

* a) The Subject is a woman who is pregnant or lactating. b) Contralateral knee has already been enrolled in this study . c) Revision knee that was previously enrolled in the study as a primary knee (ipsilateral).

  d) Subject has participated in a clinical study with an investigational product (drug or device) in the last two (2) years.

  e) Subject has had surgery on their contralateral knee within six (6) months of study enrolment or has surgery planned on their contralateral knee less than six (6) months of the study surgery.

  f) Subject is suffering from inflammatory arthritis in any joint (e.g., rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).

  g) Active local or systemic infection. h) Loss of bone or musculature, inadequate bone quality (e.g. severe osteoporosis), neuromuscular compromise or vascular deficiency at the bone site in the affected limb in sufficient degree to render the procedure unjustifiable (e.g. absence of musculoligamentous supporting structures that could lead to implant instability, joint neuropathy).

  i) Severe instability secondary to advanced loss of osteochondral structure or the absence of collateral ligament integrity.

  j) The inability to make bone cuts (e.g. inadequate bone stock) so as to assure correct component position, a firm press fit, and intimate apposition of the cut bone and prosthetic surfaces.

  k) Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.

  l) Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last five 5 years) or has a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Morris, Study Director — DePuy Synthes
Locations (15):
- United States (15):
  - Orthopaedic Specialty Institute, Irvine, California
  - Coastal Orthopedics, Bradenton, Florida
  - Florida Orthopaedic Associates, DeLand, Florida
  - University of Florida, Gainesville, Florida
  - American Hip Institute & Orthopedic Specialists, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins Orthpaedic Surgery, Baltimore, Maryland
  - Towson Orthopaedic Associates, Baltimore, Maryland
  - Rubin Institute for Advanced Orthopedics, Baltimore, Maryland
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - University of Missouri, Columbia, Missouri
  - Mercy Clinic Springfield, Ozark, Missouri
  - University Orthopaedic Associates, LLC, Somerset, New Jersey
  - Orlin & Cohen Orthopedics, Garden City, New York
  - Anderson Clinic, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
Supporting Information: Study Protocol
Time Frame: Study Protocol will be immediately available.
Access Criteria: There are no additional qualifying criteria for access to the study protocol.
URL: https://yoda.yale.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty patients were consented and enrolled. Fifty-nine subjects underwent surgery. All subjects have now been discontinued from the study.
Pre-assignment Details: Eighty patients were consented and enrolled. Fifty-nine subjects underwent surgery. All subjects have now been discontinued from the study.
Groups:
- ATTUNE Cementless Fixed Bearing: ATTUNE Cementless Femur, ATTUNE Cementless Fixed Bearing Tibial Base, ATTUNE polyethylene insert, ATTUNE Cemented Patella or not resurfaced.
Period: Overall Study
Arm/Group | ATTUNE Cementless Fixed Bearing
Started (80) | 80
Completed (0) | 0
Not Completed | 80
Not completed — Intraoperative Screen Failure | 5
Not completed — Study terminated prematurely | 71
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Eighty patients were screened and enrolled.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Time of Consent
  Years | 63.0 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of Participant
  Participants
    Female | 50
    Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of Participant
  Participants
    Hispanic or Latino | 6
    Not Hispanic or Latino | 68
    Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 51
  More than one race | 0
  Unknown or Not Reported | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.9 (6.43)

OUTCOME MEASURES:

1. Primary Outcome: One Year Functional Responder Rate of First 225 Subjects
Description: Functional Responder Rate with an Objective Performance Criteria of 85% as measured by the KOOS questionnaire for the first 225 tibia
Time Frame: through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

2. Secondary Outcome: Measure of Knees With Adverse Events
Description: This measure will assess the percentage of knees with reported AEs throughout the duration of the study.
Time Frame: Through study completion, up to 10 months
Measure: Number; unit: % of Knees with AEs
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 80
% of Knees with AEs | 13.8

3. Secondary Outcome: Mean Number of Adverse Events Per Knee for Knees With Reported AEs
Description: This measure will assess the mean number of AEs per Knee for those knees with reported AEs throughout the duration of the study.
Time Frame: Through study completion, up to 10 months
Population: 6 subjects experienced at least 1 AE
Measure: Mean (Full Range); unit: Mean Number of AEs per Knee
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 6
Mean Number of AEs per Knee | 1.83 [0.0 to 5.0]

4. Secondary Outcome: Measure of Knees With Device Deficiencies
Description: This measure will assess count of knees with various types of device deficiencies reported throughout the duration of the study.
Time Frame: Through study completion, up to 10 months
Population: There were no reported device deficiencies.
Measure: Number; unit: % of Knees with Device Deficiencies
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 59
% of Knees with Device Deficiencies | 0.0

5. Secondary Outcome: Mean Number of Device Deficiencies Per Knee
Description: This measure will assess the mean number of device deficiencies (DD) per knee reported throughout the duration of the study.
Time Frame: Through study completion, up to 10 months
Population: There were no occurrences of device deficiencies reported.
Measure: Mean (Full Range); unit: Mean # of DDs per knee
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 59
Mean # of DDs per knee | 0.0 [0.0 to 0.0]

6. Secondary Outcome: One Year Functional Responder Rate All Subjects
Description: Functional Responder Rate with an Objective Performance Criteria of 85% as measured by the KOOS questionnaire for all subjects.
Time Frame: Through study completion, up to 10 months.
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

7. Secondary Outcome: One Year Kaplan-Meier Implant Survivorship
Description: Number/rate of subjects with all implants remaining implanted at the 1 year timepoint.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

8. Secondary Outcome: Two Year Kaplan-Meier Implant Survivorship
Description: Number/rate of subjects with all implants remaining implanted at the 2- year timepoint.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

9. Secondary Outcome: Five Year Kaplan-Meier Implant Survivorship
Description: Number/rate of subjects with all implants remaining implanted at the 5- year timepoint.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

10. Secondary Outcome: 6 Week Knee Society Score
Description: Mixed outcome measure that derives a score using physician input and patient input including current symptoms, knee function, patient satisfaction and expectations.
Time Frame: Through study completion, up to 6 weeks
Population: This includes analysis for all subjects with scorable KSS forms. Not all visits yielded scorable forms. For all categories, higher values are considered better than lower values.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 42
Scores on a scale
  Alignment Subscore: Max 25 (more aligned), Min 0; Knee Alignment | 23.3 (7.54)
  Instability Subscore: Max 25 (more stable), Min 0; Stability in the Coronal and Sagittal Axis. | 24.8 (1.08)
  Joint Motion Subscore: Max 25 (more degrees of motion), Min 0; Degrees of Joint Motion. | 15.71 (2.381)
  Symptoms Subscore: Max 25 (least pain), Min 0; Patient Rating of pain with walking. | 15.5 (5.18)
  Objective Total Score: Max 100 (best), Min 0; Total Alignment, Instability, Motion, and Symptoms. | 81.45 (5.510)
  Patient Satisfaction Total Score: Max 40 (best), Min 0; Measure of Patient's Level of Satisfaction | 25.1 (7.25)
  Patient Expectation Total Score: Max 15 (best), Min 0; Patient's Expectations the Surgery | 9.7 (2.98)
  Patient Function Total Score: Max 100 (best), Min 0; Walking, Standing, and Other Activities. | 38.4 (10.9)

11. Secondary Outcome: 6 Month Knee Society Score
Description: as for outcome 10
Time Frame: Through study completion, up to 6 Months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 10
Scores on a scale
  Alignment Subscore: Max 25 (more aligned), Min 0; Knee Alignment | 25.0 (0.00)
  Instability Subscore: Max 25 (more stable), Min 0; Stability in the Coronal and Sagittal Axis. | 24.4 (1.67)
  Joint Motion Subscore: Max 25 (more degrees of motion), Min 0; Degrees of Joint Motion. | 18.87 (3.477)
  Symptoms Subscore: Max 25 (least pain), Min 0; Patient Rating of pain with walking. | 20.0 (4.36)
  Objective Total Score: Max 100 (best), Min 0; Total Alignment, Instability, Motion, and Symptoms. | 88.31 (5.367)
  Patient Satisfaction Total Score: Max 40 (best), Min 0; Patient's Level of Satisfaction | 32.4 (5.56)
  Patient Expectation Total Score: Max 15 (best), Min 0; Patient's Expectations the Surgery | 12.8 (3.01)

12. Secondary Outcome: One Year Knee Society Score
Description: Mixed outcome measure that derives a score using physician input and patient input including current symptoms, knee function, patient satisfaction and expectations. The higher the score, the better the function, satisfaction, and expectations.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint. For all categories, higher values are considered better than lower values.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

13. Secondary Outcome: Two Year Knee Society Score
Description: as for outcome 12
Time Frame: Through study completion, up to 10 months
Population: as for outcome 12
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

14. Secondary Outcome: Five Year Knee Society Score
Description: as for outcome 12
Time Frame: Through study completion, up to 10 months
Population: as for outcome 12
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

15. Secondary Outcome: Six Week Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: A knee-specific instrument that derives a score developed to assess the patients' opinion about their knee and associated problems. The scores for each dimension are calculated by summing the answers to the questions. The resulting scores are then transferred to a scale from 0 to 100 with 0 representing extreme knee problems and 100 representing no problems.
Time Frame: Through study completion, up to 6 weeks
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 41
Scores on a scale
  Pain Subscore: Max 100 (best), Min 0; Patient Pain Rating. | 60.65 (16.403)
  Symptoms Subscore: Max 100 (best), Min 0; Patient Knee Symptoms. | 57.13 (14.293)
  Activities of Daily Living Function Subscore: Max 100 (best), Min 0: Patient's ability to do ADLs. | 66.75 (14.937)
  Sports and Recreation Subscore: Max 100 (best), Min 0; Ability to do Sports and Recreation. | 26.49 (18.517)
  Quality of Life Subscore: Max 100 (best), Min 0; Patient Measure of Quality of Life. | 45.73 (16.022)

16. Secondary Outcome: Six Month Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 15
Time Frame: Through study completion, up to 6 Months
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 10
Scores on a scale
  Pain Subscore: Max 100 (best), Min 0; Patient Pain Rating. | 81.11 (20.108)
  Symptoms Subscore: Max 100 (best), Min 0; Patient Knee Symptoms. | 61.07 (9.737)
  Activities of Daily Living Function Subscore: Max 100 (best), Min 0: Patient's ability to do ADLs. | 82.50 (16.382)
  Sports and Recreation Subscore: Max 100 (best), Min 0; Ability to do Sports and Recreation. | 52.50 (23.244)
  Quality of Life Subscore: Max 100 (best), Min 0; Patient Measure of Quality of Life. | 68.96 (21.594)

17. Secondary Outcome: One Year Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 15
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

18. Secondary Outcome: Two Year Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 15
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

19. Secondary Outcome: Five Year Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 15
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

20. Secondary Outcome: Six Week Forgotten Joint Score (FJS-12)
Description: The Forgotten Joint Scores comprise measures for the assessment of joint-specific patient-reported outcome (PRO). These PRO questionnaires focus on patients' awareness of a specific joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. This may include strong sensations like pain, but also includes more subtle feelings like mild stiffness, subjective dysfunction, or any discomfort. The FJS-12 score ranges from 0 to 100, with 0 being the worst score and 100 being the best. A higher score means the patient is better able to forget about the artificial joint in daily life. So, the higher the score, the better the outcome is
Time Frame: Through study completion, up to 6 weeks
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 41
Scores on a scale | 20.07 (17.701)

21. Secondary Outcome: Six Month Forgotten Joint Score (FJS-12)
Description: as for outcome 20
Time Frame: Through study completion, up to 6 months
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 9
Scores on a scale | 49.54 (16.463)

22. Secondary Outcome: 1 Year Forgotten Joint Score (FJS-12)
Description: as for outcome 20
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

23. Secondary Outcome: Two Year Forgotten Joint Score (FJS-12)
Description: as for outcome 20
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

24. Secondary Outcome: Five Year Forgotten Joint Score (FJS-12)
Description: as for outcome 20
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

25. Secondary Outcome: Six Week EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. Scores are derived by a 5 digit code. The higher the number, the better the overall health status of the patient.
Time Frame: Through study completion, up to 6 weeks
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 40
Scores on a scale
  EQ VAS Total Health Score: Max 100 (best), Min 0; Patient's perception of their health. | 76.6 (11.81)
  EQ-5D-5L Index Value: Max 1.0 (best), Min 0.0; Measure of patient health for appraisal. | 0.7398 (0.1326)

26. Secondary Outcome: Six Month EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Through study completion, up to 6 months
Population: Analysis not completed due to early closure of the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 9
Scores on a scale
  EQ VAS Total Health Score: Max 100 (best), Min 0; Patient's perception of their health. | 85.6 (12.10)
  EQ-5D-5L Index Value: Max 1.0 (best), Min 0.0; Measure of patient health for appraisal. | 0.8780 (0.0738)

27. Secondary Outcome: One Year EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

28. Secondary Outcome: Two Year EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

29. Secondary Outcome: Five Year EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

30. Secondary Outcome: Six Month Investigator-conducted Radiographic Analysis
Description: Rate of radiolucencies and other significant radiographic findings identified by clinical investigators.
Time Frame: Through study completion, up to 6 Months
Measure: Number; unit: % of Knees with Significant Findings
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 50
% of Knees with Significant Findings
  Osteolysis | 2.0
  Radiolucency | 2.0

31. Secondary Outcome: One Year Investigator-conducted Radiographic Analysis
Description: Rate of radiolucencies and other significant radiographic findings identified by clinical investigators.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

32. Secondary Outcome: Two Year Investigator-conducted Radiographic Analysis
Description: Rate of radiolucencies and other significant radiographic findings identified by clinical investigators.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

33. Secondary Outcome: Five Year Investigator-conducted Radiographic Analysis
Description: Rate of radiolucencies and other significant radiographic findings identified by clinical investigators.
Time Frame: Through study completion, up to 10 months
Population: Data were not collected as the study terminated prior to the pre-specified analysis timepoint.
Arm/Group | ATTUNE Cementless Fixed Bearing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the preoperative visit to study closure, up to 10 months.
Description: All serious, device-related, and/or procedure-related adverse events were reported throughout the duration of the study.
Arm/Group | ATTUNE Cementless Fixed Bearing
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 6/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATTUNE Cementless Fixed Bearing (N=80)
Right Knee Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATTUNE Cementless Fixed Bearing (N=80)
Swelling on Left Ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising on Left Leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Numbness on Lateral Side (Musculoskeletal and connective tissue disorders) | 2 (2)
Limited Range of Motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pins and Needles L Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cemented the Tibial Base (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary/secondary endpoint analyses were not conducted due to early termination of the clinical study. Due to early study closure and the limited amount of post-operative clinical evidence collected during this clinical investigation, limited conclusions can be made regarding the overall safety and performance of the ATTUNE AFFIXIUM Tibial Base. Further clinical data collection and analysis are required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data collection in this study was conducted according to the Clinical Investigation Plan and all applicable regulations unless otherwise stated. Data is not anticipated to be used for publication or as the basis for future regulatory submissions except as part of routine post-market surveillance on the associated products. The database was closed without source data verification or final data cleanup. No statistical analysis of this data will occur.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT04630262/Prot_SAP_000.pdf